CLINICAL TRIAL: NCT05814861
Title: Isolation and Characterization of Blastocystis Hominis as Apotential Human Pathogen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Alzahraa Montaser Ali, Investigator, Assiut University
Other Study IDs: Blastocystis hominis isolation
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Blastocystis Hominis Infections
MeSH Terms: conditions — Blastocystis Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients presented with GIT symptoms: Fresh Stool samples will be collected in clean sterile cups from patients suffering from gastrointestinal symptoms attending Assiut University Hospitals and examined for detection of Blastocystis hominis
  Interventions: Diagnostic Test: culture and PCR
- clinically free persons undergo routine stool analysis for any reasons other than GIT complaint: Fresh Stool samples will be collected in clean sterile cups from clinically free persons under go routine stool examination for any cause other than GIT troubles and examined for detection of Blastocystis hominis
  Interventions: Diagnostic Test: culture and PCR

INTERVENTIONS:
Diagnostic Test: culture and PCR — Stool samples will be cultured inTwo media :
  A-Locke egg serum medium (LE) B- Jones' medium Then Molecular identification of Blastocystis hominis using polymerase chain reaction (PCR).

SUMMARY:
* Detection of the presence of Blastocystis hominis among outpatients presented with GIT symptoms at Assiut University Hospitals in comparison with those in control group.
* Assessment of different culture techniques for detection, and isolation of Blastocystis hominis.
* Molecular identification of Blastocystis hominis using polymerase chain reaction (PCR).

DETAILED DESCRIPTION:
Blastocystis is a genus of single-celled parasites belonging to a group of organisms that are known as the Stramenopiles . Blastocystis consists of several species, living in the gastrointestinal tracts of humans and farm animals. Many different species can infect humans and would be identified as Blastocystis hominis depending on the sequencing of the gene encoding the 18S rRNA . Among the subtypes recognized, ST1-8 could colonize humans as well as animals.

Infection with B. hominis has a worldwide distribution with infection rate reaches up to 60% in developing countries. Initially B.hominis was accepted as a harmless commensal in the intestinal tract, but recently it was implicated as a pathogen. As it able to produce a cysteine protease which breaks up the mucosal IgA antibody. B.hominis infection has been associated with several gastrointestinal symptoms, Even though most cases are asymptomatic, it is also play a significant role in some chronic gastrointestinal illnesses as irritable bowel syndrome (IBS).

Blastocystis spp. are polymorphic parasites with multiple morphological forms including vacuolar, multivacuolar, granular, ameboid, and cystic forms. At least two out of three infections may be missed during microscopic detection of B.hominis due to their polymorphic nature, and the possibility of confusion with yeast, Cyclospora spp. or fat globules. . Different studies suggested that it multiply rapidly in culture medium and considered it a sensitive method for diagnosis of B.hominis . Recently Molecular diagnosis by polymerase chain reaction (PCR) is considered the most sensitive method for the detection of B.hominis.

ELIGIBILITY:
Inclusion Criteria:

* The persons selected for the study are those who are:

  1. Suffering from any GIT manifestations, attending outpatient clinics of Internal Medicine and Tropical Medicine Departments at Assiut University Hospitals (case group)
  2. clinically free persons undergo routine stool analysis for any reasons other than GIT complaint.(control group)

Exclusion Criteria:

* We will exclude any patient who received antibiotic or anti-parasitic drugs the past 4 weeks prior to sample collection.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The persons selected for the study are those who are:
  1. Suffering from any GIT manifestations, attending outpatient clinics of Internal Medicine and Tropical Medicine Departments at Assiut University Hospitals (case group)
     * GIT manifestations such as diarrhea; (frequency ≥3 loose stool /day), either acute diarrhea (duration less than 2 weeks), or chronic diarrhea (duration more than 4 weeks), or other GIT complaints as abdominal pain, flatulence, nausea, vomiting, or weight loss.
  2. clinically free persons undergo routine stool analysis for any reasons other than GIT complaint.(control group)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
-Morphological identification of Blastocystis hominis in stool. | 1year
  Microscopic Detection of Blastocystis hominis among outpatients presented with GIT symptoms at Assiut University Hospitals .

SECONDARY OUTCOMES:
Molecular identification of Blastocystis hominis | 1 year
  Molecular identification of Blastocystis hominis using polymerase chain reaction (PCR).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A. F. Bafghi, R. Hosseini, H. R. Mollaei, and K. Barzegar, "Geno-typing and Comparison of Conventional and Molecular Diagnostic Techniques for Detection of Blastocystis on health centers in Kerman , Iran," vol. 8, no. 01, pp. 10-16, 2021..
- [Background] S M. Journal, "SOHAG MEDICAL JOURNAL Vol. 21 No.3," vol. 21, no. 3, 2017.
- [Background] M. Q. Khairuzzaman, "No Title血清及尿液特定蛋白检测在糖尿病肾病早期诊断中的意义," vol. 4, no. 1, pp. 64-75, 2016.